CLINICAL TRIAL: NCT01745796
Title: Impact of the Contamination Mode on the Clinical Evolution During Pseudomonas Aeruginosa Ventilator Acquired Pneumonia
Brief Title: Impact of the Contamination Mode on the Clinical Evolution During Pseudomonas Aeruginosa Ventilator Acquired Pneumonia (PYO GEN)
Acronym: PYO GEN
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 12SC02
Record Dates: First submitted 2012-10-08; First posted 2012-12-10 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-05

CONDITIONS: Pseudomonas Aeruginosa; Ventilation Acquired Pneumonia
Keywords: Pseudomonas Aeruginosa; Ventilated Acquired Pneumonia; Transmission modes
MeSH Terms: conditions — Pseudomonas Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — In order to achieve an antibiogram according to conventional methods and PCR genotyping Rep (DiversiLab ®) to assess the clonality of bacterial populations, there will be taken 5 different isolated colonies (possibly diluted)from each clinical sample of bronchial secretion, selected according to morphological criteria or randomly if no visible differences are noted.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intubated ICU patients

SUMMARY:
Pseudomonas aeruginosa is the main pathogen of nosocomial respiratory infections. Its increasing resistance to antibiotics requires the development of new strategies for prevention and control, demanding a better understanding of the modes of transmission and evolutionary dynamics of this bacteria. In patients under invasive mechanical ventilation, the main mode of contamination by Pseudomonas remains debated, with 3 modes of contamination (endogenous, crossed transmission between patients, or environmental origin) of varying importance, mainly depending on the endemic situation of the place of study.

The emergence of new genotyping technologies (DiversiLab) can now facilitate studies of molecular epidemiology. Thanks to the multidisciplinary collaboration and innovative techniques, the investigators wish to study the impact of the mode of contamination on the outcome of ICU patients, intubated and ventilated for more than 72 hours.

DETAILED DESCRIPTION:
The presence of environmental reservoirs can cause infections and multidrug-resistant P. aeruginosa colonization with P. aeruginosa is itself a prognostic factor, but the impact of the route of infection on the evolution of the history and future of the infectious patient is not established.

A second factor that may influence the evolution infectious is the degree of genetic heterogeneity of the bacterial population. Multiple exposure pathways could also influence the genetic diversity.

ELIGIBILITY:
Inclusion Criteria:

* Patients> 18 years
* hospitalized in the intensive care unit
* with more than 72 hours of mechanical ventilation
* Presenting a positive bacteriological sample P. aeruginosa.

Exclusion Criteria:

* Minors.
* Pregnant or lactating women.
* Patients under guardianship, under judiciary placement, or hospitalized without their consent.
* Patients not affiliated to a social security scheme.
* Long-term corticosteroid therapy (> 2mg/kg or> 1 month before the onset of established infection suspected)
* Ongoing chemotherapy, AIDS, transplant patient under immunosuppressive drugs.
* Bedridden patient or therapeutic decision at ICU arrival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients over 72 hours of intubation and mechanically ventilated
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2013-07-03; Primary Completion 2015-06-02 (Actual); Study Completion 2015-06-02 (Actual)

PRIMARY OUTCOMES:
The occurrence of unfavorable patient's outcome, depending on the mode of contamination, such as persistence, relapse or superinfection of the airways at Day 7, and mortality at Day 28 | From day 3 of intubation until the end of mechanical ventilation (an average of 28 days).

SECONDARY OUTCOMES:
Number of different clones of P. aeruginosa found in each sample analyzed for the same patient at diagnosis of colonization and VAP. | From day 3 of intubation until the end of mechanical ventilation (an average of 28 days).
  Samples of infected patients are analyzed once a week, strains are considered from different clones if their genetic homology rate is below 97%

CONTACTS AND LOCATIONS:
Locations (1):
- Medical ICU of Universitary Hospital of Grenoble, Grenoble, Isère, France